CLINICAL TRIAL: NCT05242978
Title: Acute Impact of Different Foods and Beverages on Exercise Induced Oxidative Stress and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Daniel König, Principal Investigator, University of Vienna
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2021-00743
Record Dates: First submitted 2022-01-26; First posted 2022-02-16 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2024-11

CONDITIONS: Inflammatory Response; Oxidative Stress; Oxidative Stress Induction
MeSH Terms: interventions — Nutritional Status

STUDY DESIGN:
Intervention Model Description: acute consumption of anti- and pro- inflammatory foods (n=22) and beverages (n=20) 2 hour prior to intense physical activity in healthy female subjects (in total 42 subjects)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Impact of GT, coffee, OJ, PGJ, milk, SSB on exercise induced oxidative stress&inflammation (Experimental): single consumption of one cup of green tea (GT), coffee, orange juice (OJ), pomegranate juice (PGJ), milk and sugar sweetened beverage (SSB) 2 hours prior to a 30-min- HIIT resistance circuit exercise in healthy human subjects
  Interventions: Other: Nutrition
- Impact of choc, bcc, fl-oil, blueb., r&w bread on exercise induced oxidative stress&inflammation (Experimental): single consumption of one proportion of dark chocolate (choc), broccoli (bcc), flaxseed oil, blueberries, white bread and whole grain bread (r = refined & w = whole grain) 2 hours prior to a 30-min-HIIT resistance circuit exercise in healthy human subjects
  Interventions: Other: Nutrition

INTERVENTIONS:
Other: Nutrition — acute single dose nutrition intervention

SUMMARY:
The aim of this research project is to explore the acute impact of specific foods and beverages, which have been shown to be associated with inflammatory processes, mainly in epidemiological studies, on inflammatory and oxidative stress parameters in healthy humans following a high intensity physical workout.

DETAILED DESCRIPTION:
The aim of this research project is to explore the acute impact of specific foods and beverages, which have been shown to be associated with inflammatory processes, mainly in epidemiological studies, on inflammatory and oxidative stress parameters in healthy humans following a high intensity physical workout. The choice of food will mainly be based on the food groups from the Empirical Dietary Inflammatory Index. For that purpose, forty-two healthy volunteers will be recruited to perform several interventions in order to assess the impact of different nutrient groups or single- foods on oxidative and inflammatory markers. They will be divided into two groups (beverage consumption, n=20 & plantbased foods, n=22). The intense physical activity serves to induce a physiological stress response in the body, known to be accompanied by an increase in oxidative and inflammatory stress parameters. The idea is that anti- inflammatory or antioxidant nutrients could potentially attenuate this stress response in dependence on their anti- inflammatory or antioxidant potential. The operability of this concept has already been tested. The main benefit of this approach is to get a deeper insight into short term effects of single foods or beverages on inflammatory and prooxidative processes in humans by using short term intense physical activity as a stress model. One major practical aspect of this approach is to assess dietary components with respect to their pro- or anti-inflammatory-/oxidative stress potential regarding e.g. non-communicable diseases such as type 2 diabetes, coronary heart disease or the metabolic syndrome. Furthermore, it could help to reduce inflammation or oxidative stress during or following high intense physical exercise in order to reduce the stress response during training or competition in order to enhance regeneration and to foster the training gain in sports.

ELIGIBILITY:
Inclusion Criteria:

* female human subjects
* aged 18-40 years
* no chronical diseases
* not more than 120 minutes of physical activity per week
* no regular resistance training within the past 6 months
* BMI 18.5 - 24.99 kg/m²
* body fat percentage of at least 20%
* Exclusion Criteria:
* contraindications against physical activity
* anemia
* fructose or lactose intolerance
* smoking
* medications with influence on ROS levels or inflammation
* allergy or intolerance against intervention food/beverages.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
ROS change | change from baseline to 2.5 hours
  ROS (change from baseline = after overnight fasting to post exercise (=after 2.5 hours)
IL-6 change | change from baseline to 2.5 hours
  IL-6 (change from baseline = after overnight fasting to post exercise (=after 2.5 hours)

SECONDARY OUTCOMES:
estradiol | baseline
  17-beta-estradiol
DNA damage (comet assay | change from baseline to 2.5 hours
  comet assay - wholeblood
MDA change | change from baseline to 2.5 hours
  MDA (change from baseline = after overnight fasting to post exercise (=after 2.5 hours)
hs-CRP change | change from baseline to 2.5 hours
  hs-CRP (change from baseline = after overnight fasting to post exercise (=after 2.5 hours)
FRAP | change from baseline to 2.5 hours
  Ferric Reducing Antioxidant Power Assay
Polyphenol Content | change from baseline to 2.5 hours
  Polyphenol Content Plasma
Lipidomics | change from baseline to 2.5 hours
  oxLDL
Protein Carbonyls | change from baseline to 2.5 hours
  Protein Carbonyl Assay

CONTACTS AND LOCATIONS:
Overall Officials: Markus Gassner, MSc, Principal Investigator — University Assistant; Daniel König, Univ Prof, Study Director — Professor of sports nutrition
Locations (1):
- University of Vienna, Vienna, Austria, Austria

IPD SHARING:
Plan to Share IPD: No